CLINICAL TRIAL: NCT04605055
Title: The Interplay Between Oxalate, Immunity and Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not started due to shift in research efforts and funding.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tanecia Mitchell, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300005965
Record Dates: First submitted 2020-10-12; First posted 2020-10-27 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Kidney Stone
Keywords: Oxalate
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Oxalate Diet Followed by High Oxalate Diet (Experimental): Subjects will consume a low oxalate diet for four days, with blood collections on Days 1 and 4 and 24-hour urine collections on Days 3 and 4. A ten day wash out period will follow, during which participants will consume their normal diet. After the wash out period, subjects will consume a high oxalate diet for four days, with blood and 24-hour urine collections occurring again as described previously.
  Interventions: Dietary Supplement: Low Oxalate Diet; Dietary Supplement: High Oxalate Diet
- High Oxalate Diet Followed by Low Oxalate Diet (Experimental): Subjects will consume a high oxalate diet for four days, with blood collections on Days 1 and 4 and 24-hour urine collections on Days 3 and 4. A ten day wash out period will follow, during which participants will consume their normal diet. After the wash out period, subjects will consume a low oxalate diet for four days, with blood and 24-hour urine collections occurring again as described previously.
  Interventions: Dietary Supplement: Low Oxalate Diet; Dietary Supplement: High Oxalate Diet

INTERVENTIONS:
Dietary Supplement: Low Oxalate Diet — Participants will consume a diet that is controlled in its daily contents of oxalate and calcium, and in its content of carbohydrate, fat, and protein.
Dietary Supplement: High Oxalate Diet — Participants will consume a diet that is controlled in its daily contents of oxalate and calcium, and in its content of carbohydrate, fat, and protein.

SUMMARY:
This study consists of having subjects, those with calcium oxalate kidney stones as well as healthy controls, consume low and oxalate enriched diets to investigate the role of oxalate on crystalluria (the presence of crystals in urine), immunity and infection.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Body Mass Index (BMI) between 20-30 kg/m2
* Non tobacco users or not pregnant/breast feeding/nursing
* Normal fasting blood comprehensive metabolic panel, complete blood count, C-reactive protein, and urinalysis. Must accurately collect two 24-hour urine collections within 20% of appropriate ratio of creatinine (mg)/body weight (kg) for gender
* Healthy subjects: No history of calcium oxalate kidney stones (CaOx KS) or other medical conditions
* Patients with CaOx KS: Recent stone composition greater than 50% CaOx; no uric acid or struvite stone content must be present. Must be first time or recurrent CaOx stone former (last stone event within the past 3 years)
* Willing to not consume supplements (i.e. vitamins, Ca (citrate or carbonate) and other minerals, herbal supplements, nutritional aids, and probiotics) for 2 weeks before the study and during the study
* Willing to abstain from vigorous exercise during the study as this may compromise immune function.
* Willing to consume diets provided only by the University of Alabama Center for Clinical and Translational Science Bionutrition Core. No food allergies or intolerance to any of the foods on the study menus.
* Willing to accurately collect 24-hour urine samples, and to have blood drawn throughout the study.
* If on medications for kidney stone prevention (e.g. thiazides, citrate supplementation excluding calcium citrate), patients must be on a stable dose regimen for at least 8 weeks prior to and during screening, with no changes in dosing anticipated during the study. Patients should not take allopurinol for 2 weeks prior to screening since allopurinol has anti-oxidant properties.

Exclusion Criteria:

* Failure to meet the inclusion criteria or physician refusal
* Inability to sign and read the informed consent
* Any medical, psychiatric, or social conditions that would prohibit participants from abiding to the study requirements
* BMI greater than 30 kg/m2 or less than 20 kg/m2
* Tobacco users or pregnant or breast feeding/nursing women
* Abnormal fasting blood comprehensive metabolic panel, complete blood count, C-reactive protein, and urinalysis. Inaccurate 24-hour urine collections.
* Healthy subjects: Taking medications or dietary supplements. History of kidney stones or any medical condition that could influence absorption or excretion of oxalate.
* Active illness including COVID-19, flu, common cold, fever, diarrhea, urinary tract infections or other infections 14 days before the study and throughout the study.
* Active disease including diabetes, gout, hypertension, primary hyperoxaluria, nephrotic syndrome, enteric hyperoxaluria, renal tubular acidosis, primary hyperparathyroidism, liver disease, autoimmune disorder, neurogenic bladder, urinary diversion, and bariatric surgery.
* Active malignancy or treatment for malignancy within 12 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Urinary Oxalate | Change between Baseline and Diets at 4 days
  Twenty-four hour urinary oxalate will be reported as mg/day
Crystalluria | Change between Baseline and Diets at 4 days
  Twenty-four hour crystalluria will be reported as particles/ml
Monocyte Cellular Bioenergetics | Change between Baseline and Diets at 4 days
  Cellular bioenergetics will be reported as oxygen consumption rate
Monocyte Mitochondrial Complex Activity | Change between Baseline and Diets at 4 days
  Monocyte mitochondrial complex activity will be reported as oxygen consumption rate
Monocyte Transcriptomics | Change between Baseline and Diets at 4 days
  Monocyte transcriptomics will be reported as gene expression (mRNA levels)

CONTACTS AND LOCATIONS:
Overall Officials: Tanecia Mitchell, PhD, Principal Investigator — University of Alabama at Birmingham